CLINICAL TRIAL: NCT06612567
Title: Normal Variants and Pitfalls of 18F_FDG PET/CT Imaging in Pediatric Oncology
Brief Title: Normal Variants and Pitfalls of 18F_FDG PET/CT in Pediatric Oncology
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Atef Mohamed, Dr, Assiut University
Other Study IDs: Pitfalls PET/CT In pediatric
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Pitfalls of PET Scan on Pediattic
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: PET/CT — is an imaging test that can help reveal the metabolic or biochemical function of your tissues and organs. The PET scan uses a radioactive drug called a tracer to show both typical and atypical metabolic activity. A PET scan can often detect the atypical metabolism of the tracer in diseases before the disease shows up on other imaging tests, such as computerized tomography (CT) and magnetic resonance imaging (MRI).

SUMMARY:
Detection Normal variants and pitfalls of 18_F _FDG PET/CT imaging in pediatic oncology.

DETAILED DESCRIPTION:
Although pediatric cancer is relatively rare compared with adult cancer, it is the second most common cause of death, after injury in children and adolescents. lymphoma, Leukemia, and brain cancer, account for more than half of pediatric cancers, followed by neuroblastoma, soft-tissue sarcomas, Wilms tumors, and bone tumors .

18Fluorine-fluorodeoxyglucose (18F-FDG) positron emission tomography/computed tomography (PET/CT) plays an important role, staging, restaging, response to treatment in childhood malignancies. PET-only examinations have been replaced by hybrid systems in the recent decades, where PET and CT are used together in oncology. In this imaging system, PET and CT are used together for functional data and morphological information, respectively. (2) Although 18F-FDG PET/CT is now well established as an accurate method for the staging and restaging of various cancers, it is also well recognized that many false-positive results can occur .

The normal distribution of FDG uptake in children differs from adults. Also, even though FDG is used widely in oncology, it is not tumor specific. Uptake of FDG may be seen in numerous benign conditions, including inflammation, infection, and trauma. Proper interpretation of pediatric FDG PET/CT studies requires knowledge of the normal distribution of FDG uptake in children, and an insight into the physiologic variants, benign lesions, and PET/CT related artifacts.

By understanding the potential causes of misinterpretation, we can increase the accuracy of interpretation, decrease the number of unnecessary follow-up studies and improve treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* All Pediatric Cancer patients referred to nuclear medicine unit to do 18F-FDG PET/CT study.

All patients > or = 18 years.

Exclusion Criteria:

* Severely ill patients. Patients with glucose level < 200 mg/dl.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients that will underwent PET/CT scan
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Detection normal variants and pitfalls of 18F-FDG PET/CT Imaging in Pediatric oncology that interfere in PET/CT study results and interpretation. | Baseline
  Detection normal variants and pitfalls of 18F-FDG PET/CT Imaging in Pediatric oncology that interfere in PET/CT study results and interpretation by follow up with PET/CT or other imagining or clinically

REFERENCES:
- [Background] https://doi.org/10.3389/fnume.2022.825891
- [Background] Smith CS, Schoder H, Yeung HW. Thymic extension in the superior mediastinum in patients with thymic hyperplasia: potential cause of false-positive findings on 18F-FDG PET/CT. AJR Am J Roentgenol. 2007 Jun;188(6):1716-21. doi: 10.2214/AJR.06.0552. PMID 17515398
- [Background] Bicakci N, Elli M. 18Fluorine-fluorodeoxyglucose PET/CT Imaging in Childhood Malignancies. Mol Imaging Radionucl Ther. 2021 Feb 9;30(1):18-27. doi: 10.4274/mirt.galenos.2020.64436. PMID 33586403
- [Background] Vali R, Alessio A, Balza R, Borgwardt L, Bar-Sever Z, Czachowski M, Jehanno N, Kurch L, Pandit-Taskar N, Parisi M, Piccardo A, Seghers V, Shulkin BL, Zucchetta P, Lim R. SNMMI Procedure Standard/EANM Practice Guideline on Pediatric 18F-FDG PET/CT for Oncology 1.0. J Nucl Med. 2021 Jan;62(1):99-110. doi: 10.2967/jnumed.120.254110. PMID 33334912